CLINICAL TRIAL: NCT01207674
Title: Transversal Multiaxial Evaluation and 5-year Follow-up of a Cohort of French Gamblers.
Brief Title: Transversal Multiaxial Evaluation and 5-year Follow-up of a Cohort of French Gamblers (JEU)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: MILDT (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Purpose: Other
Other Study IDs: BRD/08/09-F
Record Dates: First submitted 2010-09-22; First posted 2010-09-23 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Pathological or "at Risk" Gambling
Keywords: Pathological gambling; "at risk" gambling; gambling practice evolution; psychiatric comorbidities; gambling trajectory; cognitive distortions; ADHD; addiction; recourse to care
MeSH Terms: conditions — Gambling; Attention Deficit Disorder with Hyperactivity; Behavior, Addictive

INTERVENTIONS:
Other: Summons of patients and filling questionnaire — The study is conducted at the same time by 7 French specialised centres. The recruitment period is comprised between April 2009 and September 2011.For the first stage of the study, an initial evaluation will be performed at the time of recruitment. It consists in an individual face-to-face interview based on standardized and semi-structured questionnaires, during approximately one and half hour, and focused mainly on gambling trajectory and severity, and on psychiatric and addictive comorbidities. The evaluation is completed by a set of self-administered questionnaires focused on cognitive distortions, temperament and character, ADHD, etc.For the second stage of the study, the cohort will be re-evaluated each year, based on the same questionnaires that for initial evaluation. Each participant will be followed-up during 5 years. The study will thus end up in September 2016.

SUMMARY:
This study is divided into two stages. The first stage is a transversal study and corresponds to the recruitment of participants, which will last about two years. Three groups of gamblers will be constituted : Non-problematic gamblers (NPG), Problematic gamblers Not in Care (PGNC) and Problematic gamblers in Care (PGC).The second stage is a prospective 5-year follow-up study of the cohort (only the initial NPG and PGNC groups are concerned by the follow-up study), that consists on an annual follow-up evaluation. The main objective of the first stage of the study is to compare the characteristics of the three groups of gamblers on some socio-demographic and clinical data. These comparisons will allow us to identify, among all data, those that will be most likely to explain the evolution of the practice of gambling (appearance or resolution of a gambling problem), and recourse to specific care. These such isolated data will be tested in the second stage of the study, in order to determine those that are predictive factors of three steps of the gambling course of some gamblers : evolution of a controlled gambling practice into a problematic gambling practice, resolution of the problematic gambling practice without intervention of care, and first recourse to specific care.

ELIGIBILITY:
Inclusion Criteria:

* To be 18 to 65 years old
* To have gambled during the last year
* To gamble at least one time a year

Exclusion Criteria:

* To be under tutelage (a French protecting measure for persons with altered judgement)
* To present obvious cognitive disturbances
* To have difficulties to read and/or write in French language

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 641 (Actual)
Dates: Start 2009-04; Primary Completion 2011-11 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Number of psychiatric comorbidities | 5 years
  The 10 psychiatric comorbidities explored by the MINI are major depressive episode, (hypo)-maniac episode, 5 anxiety disorders (panic disorder ± agoraphobia, social phobia, obsessional-compulsive disorder, PTSD, generalised anxiety disorder), substance use disorders (alcohol, other psychoactive substances), psychotic disorders, and eating disorders (anorexia nervosa and bulimia).

SECONDARY OUTCOMES:
Socio-demographic data | 5 years
  gender, age, marital status, educational level, professional status, professional category, and level of income per month.
Clinical data | 5 years
  psychiatric and somatic comorbidities, personality disorders, gambling habits, diagnosis and severity of pathological gambling, level of cognitive distortions, ADHD in childhood and adulthood, temperament and character.Each of these data is measured at the initial evaluation (at time of recruitment), and then each year during the time of follow-up (5 years).

CONTACTS AND LOCATIONS:
Overall Officials: Marie GRALL BRONNEC, MD, Study Director — Nantes University Hospital
Locations (7):
- France (7):
  - Bordeaux University Hospital, Bordeaux
  - Clermont Ferrand university Hospital, Clermont-Ferrand
  - Louis Mourier hospital, Colombes
  - Marseille University Hospital, Marseille
  - Nantes University Hospital, Nantes
  - Marmottan hospital, Paris
  - Paul Brousse hospital, Villejuif

REFERENCES:
- [Derived] Guillou Landreat M, Chereau Boudet I, Perrot B, Romo L, Codina I, Magalon D, Fatseas M, Luquiens A, Brousse G, Challet-Bouju G, Grall-Bronnec M; JEU-Group. Problem and non-problem gamblers: a cross-sectional clustering study by gambling characteristics. BMJ Open. 2020 Feb 18;10(2):e030424. doi: 10.1136/bmjopen-2019-030424. PMID 32075821
- [Derived] Challet-Bouju G, Hardouin JB, Venisse JL, Romo L, Valleur M, Magalon D, Fatseas M, Chereau-Boudet I, Gorsane MA; JEU Group; Grall-Bronnec M. Study protocol: the JEU cohort study--transversal multiaxial evaluation and 5-year follow-up of a cohort of French gamblers. BMC Psychiatry. 2014 Aug 20;14:226. doi: 10.1186/s12888-014-0226-7. PMID 25141820